CLINICAL TRIAL: NCT00146081
Title: Weight Management Skills in African American Outpatients
Acronym: SHARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Shiriki K. Kumanyika, Ph.D., M.P.H., R.D., University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 704086
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2008-03-31 (Estimated); Status verified 2008-03

CONDITIONS: Obesity
Keywords: African Americans; weight control; social support
MeSH Terms: conditions — Obesity

ARMS (4):
- A (Experimental): Family Program: Participants who have identified at least 1 family member or friend to enroll in SHARE with them, who are randomly assigned to program A, are invited to bring their enrolled family member or friend (co-participant) with them to the study intervention group sessions as their supportive team member.
  Interventions: Behavioral: Weight Management
- B (Active Comparator): Coach Program: Participants who identify 1 or 2 family members or friends to enroll in SHARE with them, who are randomly assigned to program B, are invited to attend the study intervention group sessions without their enrolled family or friend (co-participants). The co-participants receive the same written materials, but act as supportive team members outside of the group sessions only. They are invited to attend special field workshops and personal counseling sessions with their co-participants.
  Interventions: Behavioral: Weight Management
- C (Experimental): Team Program: Participants who do not identify 1 or 2 family or friend co-participants, and are randomly assigned to program C, are paired with other unrelated enrollees in their group sessions as supportive team members.
  Interventions: Behavioral: Weight Management
- D (Active Comparator): Individual Program: Participants who do not identify 1 or 2 family members or friends to enroll in SHARE with them, and are randomly assigned to program D, attend group sessions as individuals.
  Interventions: Behavioral: Weight Management

INTERVENTIONS:
Behavioral: Weight Management — Participants (Index Participants) who identify 1 or 2 family members or friends (Co-Participants) to enroll with them are randomly assigned into either program A or B, and those who choose to enroll by themselves are randomly assigned to either program C or D. All Index Participants are invited to attend weekly group behavior change educational sessions; weekly in first 6 months, biweekly in next 6 months, and monthly in year 2. Co-Participants in program A are invited to attend all sessions with their Index Participant, but only the field workshops and personal counseling sessions if enrolled in program B.

SUMMARY:
Our long-term goal is to identify new insights about effective approaches to obesity management and related lifestyle changes in African Americans and about factors that enhance or limit the response to specific treatment approaches. Our primary interest is in "natural social support" from family members or friends. However, since not all individuals seeking obesity treatment desire or are able to name family members or friends to participate with them, we will also study the benefits of social support by creating a "team" condition among individuals recruited alone.

Specific aims are to:

1. Recruit overweight or obese "index" participants together with 1 or 2 family members or friend co-participants who are also overweight or obese, for enrollment in a 2 year weight loss program;
2. Conduct a randomized comparison of the effects, on weight loss and related behavioral and clinical outcomes of the index participants, of involving both index and co-participants (Group A) in the counseling program with those obtained when co-participants are not directly involved (Group B);
3. Enroll otherwise eligible index participants who do not name co-participants in a parallel 2 year weight loss study; Conduct a randomized comparison of the effects, on weight loss and related behavioral and clinical outcomes of individual participants, of creating social support teams of unrelated individuals (Group C) with those obtained when no such teams are created (Group D).

Primary hypotheses are that:

1. weight loss from 0 to 12 months and from 0 to 24 months will be significantly greater in Group A vs. Group B;
2. weight maintenance from 12 to 24 months will be significantly greater in Group A vs. Group B;
3. weight loss from 0 to 12 months and from 0 to 24 months will be significantly greater in Group C vs. Group D;
4. weight maintenance from 12 to 24 months will be significantly greater in Group C vs. Group D. Secondary analyses will compare the respective treatment and control groups on changes in diet, physical activity, and clinical CVD risk factor changes over time and will assess predictors of outcomes and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* African American Men and Women
* Ages 35-70 years
* Body Mass Index 27-54

Exclusion Criteria:

* Pregnant
* Taking Weight Altering Medication

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 344
Dates: Start 2002-08; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Weight

CONTACTS AND LOCATIONS:
Overall Officials: Shiriki K Kumanyika, PhD, MPH, RD, Principal Investigator — University of Pennsylvania
Locations (1):
- 3401 Market Street, Suite 202, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Kumanyika SK, Wadden TA, Shults J, Fassbender JE, Brown SD, Bowman MA, Brake V, West W, Frazier J, Whitt-Glover MC, Kallan MJ, Desnouee E, Wu X. Trial of family and friend support for weight loss in African American adults. Arch Intern Med. 2009 Oct 26;169(19):1795-804. doi: 10.1001/archinternmed.2009.337. PMID 19858438